CLINICAL TRIAL: NCT00571974
Title: A Combined Phase I/II Single Site Study to Determine the Safety and Efficacy of Photodynamic Therapy (PDT) Utilizing 5-aminolevulinic Acid (5-ALA) and PDT in the Treatment of Premalignant Oral and/or Oropharynx Lesions.
Brief Title: Treatment of Oral Premalignant Lesions With 5-ALA PDT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 51439
Record Dates: First submitted 2007-12-05; First posted 2007-12-12 (Estimated); Results first posted 2012-11-13 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Leukoplakia; Erythroplakia
MeSH Terms: conditions — Leukoplakia; Erythroplasia | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 1 light dose escalation (Experimental): During Phase I, to determine the maximum tolerated energy density of the Pulse Dye Laser operated at 585 nm with a pulse time of 1.5 ms (PDL-585), when used in combination with 5-aminolevulinic acid (5-ALA) applied topically to the premalignant lesion.
  The maximum tolerated energy density will be called the Maximum Tolerated Dose (MTD). Procedure: Fluorescence Diagnosis Imaging Interventions: Application of 5-ALA to lesion followed by activation with high power 585 nm pulsed dye laser (PDL-585, ScleroPLUS laser) at 6, 7 and 8 J/cm2.
  Interventions: Device: PDL-585, ScleroPLUS laser; Drug: 5-Aminolevulinic Acid (Levulan KerastickTM); Procedure: Fluorescence Diagnosis Imaging
- Phase 2 - Treatment efficacy of PDT (Experimental): Procedure: Fluorescence Diagnosis Imaging
  Interventions: Application of 5-ALA to lesion followed by activation with high power 585 nm pulsed dye laser (PDL-585, ScleroPLUS laser) at 8 J/cm2.
  Interventions: Device: PDL-585, ScleroPLUS laser; Drug: 5-Aminolevulinic Acid (Levulan KerastickTM); Procedure: Fluorescence Diagnosis Imaging

INTERVENTIONS:
Device: PDL-585, ScleroPLUS laser — PDT Treatment; emits light with 585 nm wavelength in pulses of 1.5 milliseconds in sections of 5 mm diameter to target the lesion and surrounding tissue
Drug: 5-Aminolevulinic Acid (Levulan KerastickTM) — Topically administered; incubation time 60-180 minutes; single dose (345 mg of active 5-ALA in 1.5 ml solution); soaked onto white gauze and applied to lesion, covered with sterile Xeroform gauze
  Other Names: 5-ALA
Procedure: Fluorescence Diagnosis Imaging — FD Image taken prior to PDL-585 usage

SUMMARY:
Oral leukoplakia within the mouth is a visible white patch which can develop into cancer if not treated. There is no good treatment for these lesions, apart from surgery which is associated with significant side effects and physical deformation of the treated area.

The investigators hypothesized that photodynamic therapy can be used safely and effectively to induce significant regression of oral leukoplakia.

DETAILED DESCRIPTION:
This is a combined Phase I/II non-randomized prospective study designed to determine the safety and assess the clinical efficacy of PDT in the treatment of oral leukeplekia with 5-ALA and 585-nm PDL with 1.5 ms pulse time. In the first part of the study we determined the maximum tolerated dose (MTD) of the PDL radiant exposure in combination with 5-ALA. In the second phase of the study, this dose is used to treat subjects at the MTD in order to determine the efficacy of the treatment by documenting the regression of the treated lesions.

ELIGIBILITY:
Inclusion Criteria:

* At least one grossly visible premalignant lesion (i.e. leukoplakia or erythroplakia) in the oral cavity or oropharynx, with a confirmed diagnosis of leukoplakia with or without dysplasia,measuring ≥ 10 mm in diameter.
* Informed of alternative treatment methods including watchful waiting, laser ablation, or surgical resection.
* Eligible for long-term follow-up for at least one year and be able to tolerate biopsies.
* Subject has signed an informed consent.
* Subject is between the ages of 18 - 80 years of age.
* Male or Female
* Zubrod performance status of 0 or 1 at screening. See Appendix A

Exclusion Criteria:

* Known sensitivity to porphyrins or photoactive medications - See Appendix B
* Invasive carcinoma of the lesion as demonstrated by biopsy.
* Subjects with inherited or acquired blood clotting defects
* Women who are breast feeding, have a positive (+) urine pregnancy test, or refuse to use 2 effective means of contraception during drug exposure and up to 48 hours after.
* Subjects with porphyria
* Life expectancy less than 12 months
* Inability or unwillingness of subject to give written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gal Shafirstein, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Result] Shafirstein G, Friedman A, Siegel E, Moreno M, Baumler W, Fan CY, Morehead K, Vural E, Stack BC Jr, Suen JY. Using 5-aminolevulinic acid and pulsed dye laser for photodynamic treatment of oral leukoplakia. Arch Otolaryngol Head Neck Surg. 2011 Nov;137(11):1117-23. doi: 10.1001/archoto.2011.178. PMID 22106236

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were identified in the head and neck oncology clinic and enrolled into the study within the time period of January 1, 2007 to November 18, 2009.
Pre-assignment Details: Screen failure did meet incl./excl. criteria
Groups:
- Phase I: To determine the maximum tolerated energy density of the Pulse Dye Laser operated at 585 nm with a pulse time of 1.5 ms (PDL-585), when used in combination with 5-aminolevulinic acid (5-ALA) applied topically to the premalignant lesion.
  The maximum tolerated energy density will be called the Maximum Tolerated Dose (MTD).
- Phase II: During Phase II, to assess the treatment efficacy of PDL-585 when used at the MTD in combination with 5-ALA applied topically to the premalignant lesion. Treatment efficacy will be assessed by means of the 90-day Objective Response rate observed among study subjects treated at the MTD.
Period: Phase I
Arm/Group | Phase I | Phase II
Started | 9 | 0
Completed | 9 | 0
Not Completed | 0 | 0
Period: Phase II
Arm/Group | Phase I | Phase II
Started | 0 | 21 (3 participants are from phase I)
Completed | 0 | 17
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II | Total
Number analyzed (Participants) | 11 | 18 | 29
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 80 years | 11 | 18 | 29
  >=80 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 4 | 11 | 15

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Description: The traditional 3+3 dose escalation design was employed. Three cohorts were enrolled at 3 subjects per cohort, and treated with escalating radiant exposures of 6, 7, or 8 J/cm2. In each cohort, the number of dose-limiting toxicities (DLTs) were observed. Dose escalation rules were the same as those provided by Storer 1989.
Time Frame: Day 2
Population: Three cohorts were enrolled at 3 subjects per cohort, and treated with escalating radiant exposures (laser doses) of 6, 7, or 8 J/cm2. In each cohort, the number of dose-limiting toxicities (DLTs) were observed. The highest radiant light dose attained that did not produce more than 2 DLTs was declared to be the maximum tolerated dose (MTD).
Measure: Number; unit: J/cm2
Groups:
- Phase I: Participants in the Phase I part of the study.
Arm/Group | Phase I
Number analyzed (Participants) | 9
J/cm2 | 8

2. Primary Outcome: The Objective Response Rate is the Number of Participants With Significant Response (SR), Partial Response (PR) or No Response (NR).
Description: The response rate was quantified by examination by an experienced head and neck surgeon and classified as follows: significant response (SR) was one where the lesion had greater than 75% resolution, partial response (PR) was one in which the lesion was reduced in size by at least 25%, and no response (NR) was one where the lesion was reduced by less than 25% in size.
Time Frame: Day 90
Population: The Simon two-stage minimax design with 9 subjects in the first stage and 8 subjects in the second stage, yielding 17 subjects overall.
Measure: Number; unit: participants
Groups:
- Phase II: Subjects treated with the MTD.
Arm/Group | Phase II
Number analyzed (Participants) | 17
participants
  Participants with Significant Response (SR) | 7
  Participants with Partial Response (PR) | 9
  Participants with no Response (NR) | 1
Statistical Analysis 1: Comparison: Phase II; The Simon two-stage minimax design with 9 subjects in the first stage and 8 subjects in the second stage, yielding 17 subjects overall. This design's early termination rule was ≤3/9 responses in the first stage, and its success criterion was ≥7/17 responses overall. This design had 80% power at 5% alpha to distinguish an efficacious 50% response rate from a null-hypothesis 20% response rate; Test type: Superiority or Other; p = 0.0001, One-sided exact binomial test — One-sided exact binomial test to compare the observed response rate to the 20% rate envisioned under the original null hypothesis; Because all but one subject responded to treatment, the Fisher's exact test was addedd

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Phase I | Phase II
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/21
Other Adverse Events (participants affected / at risk) | 9/9 | 2/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=9) | Phase II (N=21)
Pain (Nervous system disorders) | 2 (2) | 2 (2)
Dry mouth (General disorders) | 1 (1) | 0 (0)
Bad breath (General disorders) | 1 (1) | 0 (0)
Insomnia (General disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Swollen lip (General disorders) | 1 (1) | 0 (0)
Redness on chin (General disorders) | 1 (1) | 0 (0)
Taste altered (General disorders) | 1 (1) | 0 (0)
Burning sensation (General disorders) | 1 (1) | 0 (0)
Sensitive to cold (General disorders) | 1 (1) | 0 (0)
Sensitive (General disorders) | 1 (1) | 0
Raw (General disorders) | 1 (1) | 0
Soreness (General disorders) | 1 (1) | 0
Swelling (General disorders) | 1 (1) | 0

LIMITATIONS AND CAVEATS:
Since all but one subject responded to treatment, no correlative analysis of response with change in expression of p53 or Ki-67 was undertaken.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes